CLINICAL TRIAL: NCT05568225
Title: A Phase 2 Open-Label Study to Evaluate Etavopivat for the Treatment of Anemia in Patients With Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Etavopivat for the Treatment of Anemia in Patients With Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility assessment concluded low likelihood of the trial showing meaningful patient benefit.
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4202-ONC-203
Record Dates: First submitted 2022-09-15; First posted 2022-10-05 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Very Low Risk, Low Risk, or Intermediate Risk MDS Per IPSS-R
Keywords: Anemia; Myelodysplastic Syndromes; MDS; Pyruvate Kinase; Activator; Transfusion dependent; FT-4202; Etavopivat; IPSS-R very low risk; IPSS-R low risk; IPSS-R intermediate risk; ESA refractory; ESA intolerant; Luspatercept refractory; Luspatercept intolerant
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etavopivat 400 mg QD daily (Experimental): Non-transfusion dependent (NTD), Low transfusion burden (LTB) , and High transfusion burden (HTB) patients
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — 400 mg once daily
  Other Names: FT-4202

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of etavopivat (FT-4202) for the treatment of anemia in adult patients with very low risk, low risk, or intermediate risk MDS.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient has provided documented informed consent; the informed consent form (ICF) must be reviewed and signed by each patient prior to any study-related assessments/procedures being conducted.
2. Age ≥ 18 years at time of first dose.
3. Patients, if female and of childbearing potential, must agree to use acceptable methods of contraception and agree not to donate ova from study start to 90 days after the last dose of study drug, and who if male are willing to use acceptable methods of contraception and agree not to donate sperm, from study start to 90 days after the last dose of study drug.
4. Documented diagnosis of idiopathic/de novo MDS according to World Health Organization (WHO) classification that meets the IPSS-R classification of very low, low, or intermediate risk disease, and:

   * < 5% blasts in bone marrow based on local pathology review
   * < Intermediate risk cytogenetic abnormalities per IPSS-R
5. Anemia defined as:

   * Non-transfusion dependent (NTD): Subjects with mean Hb concentration < 10.0 g/dL of 2 measurements (1 performed within 3 days prior to Day 1 and the other performed 7 to 28 days prior to Day 1, not influenced by RBC transfusion within 7 days of measurement) and < 3 RBC transfusions for anemia in the prior 16 weeks before Day 1 of etavopivat dosing

   OR
   * Transfusion dependent (TD): Subjects having received ≥ 3 units of RBCs for the treatment of anemia within 16 weeks prior to Day 1
6. Serum erythropoietin level > 200 U/L, OR, if ≤ 200 U/L, subject is non-responsive, refractory, or intolerant to erythropoiesis-stimulating agents, or erythropoiesis-stimulating agents are contraindicated or unavailable.
7. ECOG performance status of ≤ 2
8. Subject is non-responsive, refractory, or intolerant to luspatercept, or luspatercept is contraindicated or not indicated.
9. No alternative treatment options are available and/or appropriate for the subject, at the discretion of the investigator.
10. Patient is willing and able to adhere to the study visit schedule and other protocol requirements

EXCLUSION CRITERIA:

[MDS History]

1. MDS associated with del 5q cytogenetic abnormality and known TP53 abnormality
2. Therapy-associated MDS (eg. t-MDS) that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases
3. Known history of acute myeloid leukemia (AML)

   [Medical Conditions]
4. Female who is breast feeding or pregnant
5. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding
6. Absolute neutrophil count < 500/µL (0.5 x 10^9/L)
7. Platelet count < 50,000/µL (50 x 10^9/L) without transfusion support within 2 weeks
8. Hepatic dysfunction characterized by:

   * Alanine aminotransferase (ALT) > 5.0 × upper limit of normal (ULN)
   * Total bilirubin > 3.0 × ULN
   * History of cirrhosis
9. Severe renal dysfunction (estimated glomerular filtration rate at the Screening visit; calculated by the local laboratory < 30 mL/min/1.73 m^2 ) or on chronic dialysis.
10. Patients with clinically significant and active bacterial, fungal, parasitic, or viral infection.

    * Patients with acute bacterial, fungal, parasitic, or viral infection requiring systemic therapy should delay Screening/ enrollment until active therapy has been completed.
    * Patients with acute viral infections without available therapies (eg, coronavirus disease 2019 [COVID-19]) should delay Screening/ enrollment until the acute infection has resolved.

    Note: Infection prophylaxis is allowed.
11. Known human immunodeficiency virus (HIV) positivity
12. Active infection with hepatitis B virus (hepatitis B surface antigen [HepBsAg] and hepatitis B core antibody [HepBcAb] positive)
13. Active hepatitis C infection
14. History of malignancy, other than MDS, within the past 2 years prior to treatment Day 1 requiring systemic chemotherapy and/or radiation.

    * Patients with malignancy considered surgically cured are eligible (eg, non-melanoma skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of the breast)
    * Patients with incidental histologic findings of prostate cancer (T1a or T1b) are eligible
15. History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

    * Unstable angina pectoris or myocardial infarction or elective coronary intervention
    * Heart disease, heart failure as classified by the New York Heart Association classification 3 or higher, or significant arrhythmia requiring treatment,
    * Pulmonary fibrosis or pulmonary hypertension which are clinically significant ie, ≥ Grade 3 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (or higher)
16. Uncontrolled hypertension, defined as repeated elevation of diastolic blood pressure ≥ 100 mmHg despite adequate treatment
17. Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable).

    [Prior/Concomitant Therapy]
18. Prior treatment with azacitidine (injectable or oral) or decitabine
19. Use of erythropoietin, other hematopoietic growth factor treatment or lenalidomide within 30 days of starting study treatment or anticipated need for such agents during the study.
20. Prior use of luspatercept:

    * NTD patients must not have received luspatercept within 30 days prior to Day 1 treatment
    * TD patients must not have received luspatercept within 16 weeks prior to Day 1 treatment
21. Receiving or use of concomitant medications that are strong inducers of cytochrome P450 (CYP)3A4/5 (see Appendix F) within 2 weeks of starting study treatment or anticipated need for such agents during the study.
22. Prior allogeneic or autologous stem cell transplant
23. Initiation of a new chelation therapy within 3 months before the first dose of study treatment.

    [Prior/Concurrent Clinical Study Experience]
24. Participated in another clinical trial of an investigational agent (or medical device) within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational agent (or medical device).

    [Other Exclusions]
25. Medical, psychological, or behavioral conditions, which, in the opinion of the Investigator, may preclude safe participation, confound study interpretation, interfere with compliance, or preclude informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), MD, Study Director — Novo Nordisk A/S
Locations (18):
- United States (8):
  - University of Miami Hospital and Clinics, Miami, Florida
  - Ocala Oncology, Ocala, Florida
  - Cedars-Sinai Medical Center, Plainsboro, New Jersey
  - Northwell Health, Plainsboro, New Jersey
  - Northwestern Memorial Hospital, Plainsboro, New Jersey
  - The Ohio State University Medical Center, Plainsboro, New Jersey
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
- University of British Columbia - St. Paul's Hospital, Vancouver, British Columbia, Canada
- France (4):
  - Nice University Hospital - Hôpital de l'Archet, Route de Saint-Antoine, Nice
  - Hopital Saint Louis, Paris
  - Master centre for France, Paris La Défense
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-1, Pessac
- Germany (5):
  - Universitoetsklinikum Heidelberg, Heidelberg
  - Charite Universitätsmedizin Berlin, Mainz
  - Universitätsklinikum Leipzig, Klinik und Poliklinik, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Universitoetsklinikum Halle (Saale), Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 10 sites in 4 countries.
Pre-assignment Details: The study was planned for 58 weeks, including 6 weeks for screening, 24 weeks for treatment, 24 weeks for extension, and 4 weeks for follow-up. It was terminated early after meeting a predefined quality tolerance limit (QTL). Of the 45 participants targeted, only 24 were screened, and 17 were enrolled into three groups: Non-transfusion dependent (NTD) N=3, Low transfusion burden (LTB) N=5, and High transfusion burden (HTB) N=9. Each participant received 400 mg of etavopivat daily.
Groups:
- Non-transfusion Dependent: Non transfusion dependent participants who had received less than equal to <= 2 RBC transfusions for anaemia within the prior 16 weeks, orally received 400 mg of etavopivat once daily for up to 48 weeks.
- Low Transfusion Burden: Low transfusion burden participants who had received 3 to 7 RBC transfusions for anaemia within the prior 16 weeks, orally received 400 mg of etavopivat once daily for up to 48 weeks.
- High Transfusion Burden: High transfusion burden participants who had received greater than equal >= 8 RBC transfusions for anaemia within the prior 16 weeks, orally received 400 mg of etavopivat once daily for up to 48 weeks.
Period: Primary Treatment Period
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Started | 3 | 5 | 9
Efficacy Evaluable Set (EES) | 1 | 2 | 4
Safety Population | 3 | 5 | 9
Full Analysis Set (FAS) | 3 | 5 | 9
Pharmacokinetic (PK) Set | 3 | 5 | 9
Completed | 1 | 2 | 4
Not Completed | 2 | 3 | 5
Not completed — Termination of the study by the Sponsor | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Disease progression | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal of conset | 1 | 0 | 4
Not completed — Adverse Event | 1 | 0 | 0
Period: Extension Treatment Period
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Started | 1 | 2 | 4
Completed | 1 | 2 | 1
Not Completed | 0 | 0 | 3
Not completed — Termination of the study by the Sponsor | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS included all participants who signed the informed consent and received at least 1 dose of etavopivat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden | Total
Number analyzed (Participants) | 3 | 5 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.3 (5.69) | 80.2 (3.49) | 71.2 (8.11) | 74.9 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 3 | 4 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 4 | 7 | 14
  Race: Not reported | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 3 | 4 | 6 | 13
  Ethnicity: Hispanic or Latino | 0 | 1 | 1 | 2
  Ethnicity: Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hematologic Improvement- Erythroid (HI-E) Response for >=8 Weeks Within 24 Weeks of Etavopivat Treatment
Description: This outcome measure reported on the combined incidence of NTD, LTB and HTB in terms of (HI-E) response for >=8 weeks duration in participants with myelodysplastic syndromes (MDS) within 24 weeks. The participants were allocated to the following arms which were defined as: 1) NTD: >=1.5 grams per deciliter (g/dL) increase in haemoglobin (Hb) from baseline maintained >=8 consecutive weeks and no transfusion of RBC units for anemia over a continuous 8-week treatment period; 2) LTB: absence of any transfusion for >=8 consecutive weeks; and 3) HTB: reduction by >=50 percent (%) of RBC units for >=8 consecutive weeks.
Time Frame: From Baseline to Week 24
Population: EES: All participants in the FAS who have completed the week 24 response visit and who have a baseline record of the primary endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 1 | 2 | 4
Percentage of participants | 0 | 50 | 25

2. Secondary Outcome: Percentage of Participants With Hematologic Improvement-Erythroid (HI-E) Response for =>8 Weeks Within 16 and 48 Weeks of Etavopivat
Description: This outcome measure focused on the combined incidence of NTD, LTB and HTB participants, evaluating HI-E lasting =>8 weeks in individuals with MDS within 16 weeks and 48 weeks. Participant's response were defined as follows: 1) NTD: an increase of =>1.5 g/dL in Hb maintained for =>8 consecutive weeks without any RBC transfusions for anemia; 2) LTB: no transfusions over =>8 consecutive weeks; and 3) HTB: a reduction of =>50% in RBC units for =>8 consecutive weeks.
Time Frame: 48 weeks
Population: FAS: All participants who signed the informed consent and received at least 1 dose of etavopivat. Data for this outcome is not analyzed due to early study termination and have been excluded from planned analyses as prespecified in statistical analysis plan (SAP).
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Hematologic Improvement- Erythroid (HI-E) Response for =>16 Weeks Within 24 and 48 Weeks of Etavopivat
Description: This outcome measure focused on the combined incidence of NDT, LTB and HTB participants, evaluating HI-E response lasting =>16 weeks in individuals with MDS within 24 weeks and 48 weeks. Participant's response were defined as follows: 1) NTD: an increase of =>1.5 g/dL in Hb maintained for =>16 consecutive weeks without any RBC transfusions for anemia; 2) LTB: no transfusions over =>16 consecutive weeks; and 3) HTB: a reduction of =>50% in RBC units for =>16 consecutive weeks.
Time Frame: 48 weeks
Population: FAS: All participants who signed the informed consent and received at least 1 dose of etavopivat. Data for this outcome is not analyzed due to early study termination and have been excluded from planned analyses as prespecified in SAP.
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of All Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Related to Etavopivat
Description: This outcome measures the total number of AEs and SAEs in participants, including AEs related to etavopivat. AEs are any unfavorable medical occurrences in participants taking the medicinal product, regardless of causality. They include new or worsening symptoms, abnormal lab findings, and exacerbations of existing conditions, documented from the first dose through 28 days after the last dose. SAEs are severe AEs that result in death, are life-threatening, require hospitalization, lead to significant disability, or involve congenital anomalies. Important medical events posing risks to the participants are also classified as SAEs. Treatment Emergent Adverse Events (TEAEs) are AEs occurring after treatment initiation, aiding in the safety assessment of etavopivat. TEAEs will be considered drug-related if assessed by the Investigator as possibly related or related, or if relationship is missing.
Time Frame: From baseline up to 48 weeks
Population: Safety population includes all participants who received at least one dose of etavopivat (including partial dosing).
Measure: Number; unit: Events
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 3 | 5 | 9
Events
  AE | 33 | 33 | 54
  SAE | 1 | 0 | 6
  AEs related to etavopivat | 0 | 0 | 1
  AEs possibly related etavopivat | 8 | 3 | 6

5. Secondary Outcome: Number of Premature Discontinuations, Dose Interruptions, and Dose Reductions
Description: The outcome measures the total number of premature discontinuations, dose interruptions and dose reductions. Premature discontinuation was defined as any discontinuation prior to week 48. A dose interruption is a temporary halt in treatment due to an AE, while a dose reduction involves lowering the dosage of the drug when AEs occur. If a participant tolerates a reduced dose for 14 days, a rechallenge with the original dose may occur after a clinic visit, but any new Grade 3 or higher AEs require treatment discontinuation and consultation with the Global Medical Monitor before resuming.
Time Frame: Within 48 weeks
Population: Safety population included all participants who receive at least one dose of etavopivat (including partial dosing).
Measure: Number; unit: Events
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 3 | 5 | 9
Events
  Premature discontinuations | 1 | 0 | 0
  Dose interruptions | 0 | 0 | 2
  Dose reductions | 0 | 0 | 0

6. Secondary Outcome: Overall Response Rate
Description: The Overall Response Rate (ORR) is defined as the percentage of participants who achieve a predefined level of response according to the 2006 International Working Group (IWG) criteria, assessed at each scheduled evaluation.
Time Frame: Up to 48 weeks
Population: Data for this outcome is not analyzed due to early study termination and have been excluded from planned analyses as prespecified in SAP.
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Duration of Response
Description: This outcome measure reported duration of response which was defined as duration of response will be summarized with quantiles based on product limit estimates (ie, Kaplan-Meier). Duration of response is defined as the time from date of first known incidence of a 2006 IWG criteria response to the most recent date that the 2006 IWG (International Working Group) criteria is not met following the initial response. If the participant has met IWG criteria throughout the period following the initial response, the participant will be censored at the latest date of end of study, loss to follow-up, or death.
Time Frame: Up to 48 weeks
Population: as for outcome 6
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Reduction in RBC Transfusions for >=8 Weeks in Participants With LTB or HTB at Study Entry
Description: This outcome measure reports reduction in RBC transfusion by 8-week interval in participants with LTB and HTB.
Time Frame: Up to 48 weeks
Population: EES: All participants in the FAS who have completed the week 24 response visit and who have a baseline record of the primary endpoint. n (number analysed) = Participants with available data for a specified category.
Measure: Mean (Standard Deviation); unit: Total RBS units
Arm/Group | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 2 | 4
Total RBS units
  Week 1-8 | 3.0 (2.83) | 5.8 (2.63)
  Week 9-16 | 2.5 (2.12) | 6.3 (1.71)
  Week 17-24 | 3.5 (2.12) | 7.5 (3.00)
  Week 25-32: number analyzed (Participants) | 2 | 3
  Week 25-32 | 5.5 (0.71) | 7.3 (1.15)
  Week 33-40: number analyzed (Participants) | 2 | 3
  Week 33-40 | 5.0 (4.24) | 6.7 (1.15)
  Week 41-48: number analyzed (Participants) | 2 | 2
  Week 41-48 | 4.5 (2.12) | 7.5 (2.12)

9. Secondary Outcome: Percent Change From Baseline in RBC Transfusion Independence for =>8 Weeks in Participants With LTB or HTB at Study Entry
Description: This outcome measure is percent change in RBC transfusion by 8-week interval in participants with LTB and HTB. Percent reduction from baseline in RBC transfusion burden is defined as -100×(Total RBC Units Transfused During Interval)/(Baseline RBC Units Transfused Per 8 Weeks).
Time Frame: Up to 48 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change of total RBC units
Arm/Group | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 2 | 4
Percent change of total RBC units
  Week 1-8 | -20.83 (64.818) | 68.75 (156.994)
  Week 9-16 | -33.33 (47.140) | 68.75 (98.219)
  Week 17-24 | -4.17 (41.248) | 120.83 (191.183)
  Week 25-32: number analyzed (Participants) | 2 | 3
  Week 25-32 | 58.33 (11.785) | 127.78 (149.381)
  Week 33-40: number analyzed (Participants) | 2 | 3
  Week 33-40 | 33.33 (94.281) | 94.44 (91.793)
  Week 41-48: number analyzed (Participants) | 2 | 2
  Week 41-48 | 25.00 (35.355) | 50.00 (0)

10. Secondary Outcome: Change From Baseline in Neutrophils and/or Platelets Counts
Description: This outcome measure reports the change from baseline in neutrophils and/or platelets counts from baseline to week 48
Time Frame: Baseline (week 0), week 48
Population: The Safety Set includes all participants who receive at least one dose of etavopivat (including partial dosing). Here, n (number analysed) = Participants with available data for a specified category.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 3 | 5 | 9
10^9 cells per liter
  Neutrophils: number analyzed (Participants) | 1 | 2 | 1
  Neutrophils | -3.200 (NA) — The standard deviation was not evaluable as data was available for only 1 participant. | -0.950 (0.0707) | -0.100 (NA) — The standard deviation was not evaluable as data was available for only 1 participant.
  Platelets counts: number analyzed (Participants) | 1 | 2 | 1
  Platelets counts | 43.0 (NA) — The standard deviation was not evaluable as data was available for only 1 participant. | -51.0 (205.06) | -8.0 (NA) — The standard deviation was not evaluable as data was available for only 1 participant.

11. Secondary Outcome: Decrease in Ferritin and Transferrin Saturation (TSAT)
Description: This outcome measure were to report decrease in ferritin and TSAT from baseline to Week 48.
Time Frame: Up to 48 weeks
Population: as for outcome 6
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Decrease in Iron Chelation Therapy
Description: This outcome measure were to report decrease of Iron chelation therapy and will be recorded at Screening and on an ongoing basis throughout the study.
Time Frame: up to 48 weeks
Population: as for outcome 6
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from first dose to date of death. If the participant was alive at last contact, the end date will be censored at the latest of either end of study, loss to follow-up, or study discontinuation.
Time Frame: Within 48 weeks
Population: as for outcome 6
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Etavopivat Plasma Concentrations
Description: This outcome measure reported Etavopivat plasma concentrations in order to assess the PK properties of etavopivat in participants with MDS. PK parameters included but not limited to were: Time to maximum observed plasma concentration, area under the plasma concentration-time curve from time zero until the last quantifiable time point (AUC0-last), from time zero to infinity (AUC0-inf), for a dosing interval (AUCtau/AUC0-24).) However due to early termination of the study, the PK parameters were not assessed and only the plasma concentrations could be assessed.
Time Frame: Weeks 1 and 4 pre-dose, post-dose 1, 2, 4, 6 hours.Week 2 and EOT (week 48):pre-dose, post-dose 1, 2 hours
Population: The PK set includes all safety set participants who have at least one evaluable concentration for etavopivat at a scheduled PK time point after the start of dosing. Here, n (number analysed) = Participants with available data for a specified category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 3 | 5 | 9
ng/mL
  Week 1 predose: number analyzed (Participants) | 3 | 4 | 9
  Week 1 predose | 0 (0) | 0 (0) | 0 (0)
  Week 1 post-dose 1 hour | 379.77 (292.748) | 904.80 (521.000) | 1016.78 (794.503)
  Week 1 post-dose 2 hour | 751.67 (393.465) | 579.60 (403.593) | 519.11 (273.776)
  Week 1 post-dose 4 hour: number analyzed (Participants) | 2 | 5 | 9
  Week 1 post-dose 4 hour | 274.50 (86.974) | 203.80 (134.884) | 165.16 (64.895)
  Week 1 post-dose 6 hour: number analyzed (Participants) | 1 | 5 | 7
  Week 1 post-dose 6 hour | 63.50 (NA) — The standard deviation was not evaluable as data was available for only 1 participant. | 101.02 (67.693) | 83.74 (40.170)
  Week 2 pre-dose: number analyzed (Participants) | 3 | 4 | 9
  Week 2 pre-dose | 27.20 (17.843) | 19.08 (9.037) | 19.20 (12.240)
  Week 2 post-dose 1 hour | 1156.00 (371.198) | 899.40 (442.555) | 1076.44 (693.907)
  Week 2 post-dose 2 hour: number analyzed (Participants) | 3 | 4 | 9
  Week 2 post-dose 2 hour | 927.00 (310.140) | 1024.00 (530.102) | 661.78 (392.238)
  Week 4 predose: number analyzed (Participants) | 2 | 5 | 9
  Week 4 predose | 17.04 (11.540) | 24.34 (23.333) | 20.26 (9.289)
  Week 4 post-dose 1 hour: number analyzed (Participants) | 2 | 4 | 9
  Week 4 post-dose 1 hour | 1050.00 (28.284) | 386.90 (214.249) | 913.20 (1013.207)
  Week 4 post-dose 2 hour: number analyzed (Participants) | 2 | 5 | 9
  Week 4 post-dose 2 hour | 526.00 (134.350) | 453.40 (179.140) | 678.49 (379.918)
  Week 4 post-dose 4 hour: number analyzed (Participants) | 2 | 4 | 9
  Week 4 post-dose 4 hour | 151.50 (12.021) | 383.73 (261.103) | 297.90 (282.646)
  Week 4 post-dose 6 hour: number analyzed (Participants) | 2 | 3 | 9
  Week 4 post-dose 6 hour | 60.75 (11.526) | 148.13 (113.650) | 121.34 (115.306)
  End of treatment pre-dose: number analyzed (Participants) | 0 | 2 | 1
  End of treatment pre-dose |  | 21.60 (5.798) | 24.20 (NA) — The standard deviation was not evaluable as data was available for only 1 participant.
  End of treatment post-dose 1 hours: number analyzed (Participants) | 0 | 1 | 1
  End of treatment post-dose 1 hours |  | 1620.00 (NA) — The standard deviation was not evaluable as data was available for only 1 participant. | 1680.00 (NA) — The standard deviation was not evaluable as data was available for only 1 participant.
  End of treatment post-dose 2 hours: number analyzed (Participants) | 0 | 1 | 1
  End of treatment post-dose 2 hours |  | 571.00 (NA) — The standard deviation was not evaluable as data was available for only 1 participant. | 815.00 (NA) — The standard deviation was not evaluable as data was available for only 1 participant.

15. Secondary Outcome: RBC 2,3-diphosphoglycerate (2,3-DPG) and Adenosine Triphosphate (ATP) Levels Over Time
Description: Etavopivat plasma concentrations were collected in order to assess the pharmacodynamic (PD) properties of etavopivat in participants with MDS.
Time Frame: Within 48 weeks
Population: as for outcome 6
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: All presented AEs are treatment emergent AEs (TEAE). TEAE is defined as any adverse event that emerges or worsens in the period from first dose of study drug to 28 days after the last dose of study drug. Safety population includes all participants who receive at least one dose of etavopivat (including partial dosing).
Arm/Group | Non-transfusion Dependent | Low Transfusion Burden | High Transfusion Burden
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/5 | 3/9
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-transfusion Dependent (N=3) | Low Transfusion Burden (N=5) | High Transfusion Burden (N=9)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-transfusion Dependent (N=3) | Low Transfusion Burden (N=5) | High Transfusion Burden (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemosiderosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (3)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (10) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (4) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The futility assessment concluded low likelihood of the trial showing meaningful participant benefit. The decision was based on a predefined QTL that required 5 or more participants to complete 16 weeks of treatment or not having 8 or more consecutive weeks of primary endpoint data. However 7 participants did not fulfill this requirement, leading to the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT05568225/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT05568225/SAP_001.pdf